CLINICAL TRIAL: NCT06913465
Title: The Impact of Hypothyroidism on Tear Production and Dry Eye Symptoms: Implications for Optometric Care
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/801
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational cross-sectional study will assess the impact of hypothyroidism on tear production and tear film stability. Conducted at DHQ Hospital dera ghazi khan over six months, the study will recruit 71 participants aged 20-60 years using a non-probability convenience sampling method. Patients with confirmed hypothyroidism will undergo tear assessment through the Schirmer I test, Tear Breakup Time (TBUT) test, and Ocular Surface Disease Index (OSDI) questionnaire. The Schirmer test will measure tear production, while TBUT will assess tear film stability.

DETAILED DESCRIPTION:
Ocular surface staining and tear osmolarity will further evaluate ocular health. Patients with systemic conditions affecting tear production, such as diabetes or rheumatoid arthritis, will be excluded. The collected data will be analyzed to determine the relationship between hypothyroidism and dry eye symptoms, aiding in better management of ocular health in hypothyroid patients. The study aims to provide valuable insights into the association between thyroid dysfunction and tear film abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-60 years.
* Confirmed diagnosis of hypothyroidism with thyroid function tests.
* No prior history of ocular surgery or significant ocular pathology.

Exclusion Criteria:

* Use of systemic medications affecting tear production (e.g., antihistamines, diuretics).
* Other systemic conditions (e.g., diabetes, rheumatoid arthritis).
* Pregnancy or lactation

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This observational cross-sectional study will assess the impact of hypothyroidism on tear production and tear film stability. Conducted at DHQ Hospital dera ghazi khan over six months, the study will recruit 71 participants aged 20-60 years using a non-probability convenience sampling method. Patients with confirmed hypothyroidism will undergo tear assessment through the Schirmer I test, Tear Breakup Time (TBUT) test, and Ocular Surface Disease Index (OSDI)
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
The Ocular Surface Disease Index (OSDI) | 12 Months
  The Ocular Surface Disease Index (OSDI) is a 12-question questionnaire used to assess the severity of dry eye symptoms and their impact on vision-related function, scored on a scale of 0 to 100, with higher scores indicating greater disability.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - DHQ Hospital, Dera Ghazi Khan, Punjab Province
  - CENUM Center Mayo Hospital Rd, Anarkali Bazaar, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No